CLINICAL TRIAL: NCT02233426
Title: Do Hypertonic Solutions Have an Impact on Nasal Eosinophilia in Allergic Rhinitis Patients?
Brief Title: Effect of Hypertonic Solutions on Allergic Rhinitis Patients
Acronym: hypertonic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Zafer Ciftci, Assist. Prof., M.D., Namik Kemal University
Other Study IDs: NKU-001
Record Dates: First submitted 2014-08-29; First posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Allergic Rhinitis
Keywords: allergic rhinitis; nasal steroid; hypertonic saline; eosinophil; symptom score
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the effectivity of using hypertonic nasal solutions alone on the symptom scores and nasal eosinophil levels of allergic rhinitis patients, retrospectively.

DETAILED DESCRIPTION:
The medical records of the patients who admitted to outpatient clinic of otorhinolaryngology department of a tertiary referral center were retrospectively investigated. The symptom scores and nasal eosinophil levels of the patients were recorded. Patients using hypertonic solutions alone or steroid nasal spray alone were compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with positive Prick's test to at least one allergen and diagnosed as having allergic rhinitis were included
* Patients who used hypertonic nasal solution alone for at least one month were included as sthe study group
* Patients who used nasal steroid spray alone or at least one month were included as sthe study group

Exclusion Criteria:

* Patients with a history of asthma, urticeria, eczama, diabetes mellitus, hypertension, COPD and other systemic diseases were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical records of patients who admitted to the outpatient clinic of a tertiary referral center was enrolled.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-09; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
The number of eosinophils in nasal secretions | The number of eosinophils in nasal secretions that was counted before the therapy and after the first month of therapy would be recorded

SECONDARY OUTCOMES:
Sinonasal Outcome Test (SNOT-22) questionairre scores | SNOT-22 scores obtained before the treatment and after the first month of treatment would be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Zafer Ciftci, Assist. Prof, Principal Investigator — Namik Kemal University
Locations (1):
- Namik Kemal University, Department of Otorhinolaryngology, Tekirdağ, Turkey (Türkiye)